CLINICAL TRIAL: NCT04880694
Title: A Randomized, Open-Label, Multi-Centre, Phase 2a Study to Evaluate the Safety and Effect of STC3141 Continuous Infusion in Subjects With Severe Corona Virus Disease 2019（COVID-19）Pneumonia
Brief Title: A Study to Evaluate the Safety and Effect of STC3141 Continuous Infusion in Subjects With Severe Corona Virus Disease 2019（COVID-19）Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grand Medical Pty Ltd. (Industry)
Collaborators: Trium Clinical Consulting (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPHIP-0202; 2021-000399-12 (EudraCT Number)
Record Dates: First submitted 2021-04-25; First posted 2021-05-11 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2021-06

CONDITIONS: Severe COVID-19 Pneumonia
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — STC3141

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to three cohorts in a 2:2:1 ratio to receive continuous infusion of STC3141 either at rate 58.3mg/hr or 87.5mg/hr up to 3 days (72hours), or to receive appropriate standard of care. All subjects in STC3141 treatment groups will also receive standard of care for their conditions as background treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: STC3141 58.3mg/hr (Experimental): Drug: STC3141 Continuous infusion of STC3141 at rate 58.3mg/hr up to 3 days (72 hours) N=10
  Interventions: Drug: STC3141
- Cohort 2: STC3141 87.5mg/hr (Experimental): Drug: STC3141 Continuous infusion of STC3141 at rate 87.5mg/hr up to 3 days (72 hours) N=10
  Interventions: Drug: STC3141
- Cohort 3: Comparator (No Intervention): Only to receive appropriate standard of care N=5

INTERVENTIONS:
Drug: STC3141 — To receive continuous infusion of STC3141 at rate 58.3mg/hr up to 3 days (72hours).
  Also to receive appropriate standard of care.
  Arms: Cohort 1: STC3141 58.3mg/hr
Drug: STC3141 — To receive continuous infusion of STC3141 at rate 87.5mg/hr up to 3 days (72hours).
  Also to receive appropriate standard of care.
  Arms: Cohort 2: STC3141 87.5mg/hr

SUMMARY:
The study is a Randomized, Open-Label, Multi-Centre, Phase 2a Study to Evaluate the Safety and Effect of STC3141 Continuous Infusion in Subjects with Severe Corona Virus Disease 2019（COVID-19）Pneumonia.

DETAILED DESCRIPTION:
Pneumonia is the most frequent and serious complication of Corona Virus Disease 2019（COVID-19）, a disease that results from severe acute respiratory syndrome coronavirus 2（SARS-CoV-2）infection with a so-called "cytokine storm", characterized by the plasma increase of many cytokines that produce long-term damage and fibrosis of lung tissue. Therefore, the development of novel therapeutic strategies to target at neutrophils associated NETs/histones may reduce the overall disease mortality rate of COVID-19.

STC3141 is a novel investigational product that can neutralize NETs/histone via charge-charge interaction. STC3141 was found to be well-tolerated in short infusions (2 hours) and continuous long-term infusions (72 hours) in healthy volunteers.

A randomized, multi-centre, phase 2a study in 25 severe COVID-19 pneumonia subjects who require hospitalization, is designed to evaluate the safety and the preliminary effect of STC3141 in this population where the treatment will be tested for the first time.

Subjects will be randomized to three cohorts in a 2:2:1 ratio to receive continuous infusion of STC3141 either at rate 58.3mg/hr or 87.5mg/hr up to 3 days (72hours), or to receive appropriate standard of care. All subjects in STC3141 treatment groups will also receive standard of care for their conditions as background treatment.

The primary objective of the study is to evaluate the safety of STC3141 in subjects with severe COVID-19 pneumonia.The secondary objective is to evaluate the preliminary effects of STC3141 in the treatment of subjects with severe COVID-19 pneumonia.As an exploratory objective, the change in biomarkers from baseline following STC3141 treatment in subjects with severe COVID-19 pneumonia will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females who are 18 years or older (inclusive).
2. Signed informed consent. Subjects are to provide informed consent prior to any study procedures being performed. Consent can be oral if a written consent cannot be expressed. Where it is not practicable to approach a subject highly dependent on medical care, or the subject is not capable of making such a decision, consent will be sought from the legal representative of the subject. Subjects enrolled in the study based on consent by the legal representative will be given the opportunity to provide written confirmatory consent when and if they become able to do so. If the subject declines to confirm consent, they will be withdrawn from the study at the point where they decline consent.
3. Virological diagnosis of severe acute respiratory syndrome coronavirus 2（SARS-CoV-2）infection (documentation of real-time polymerase chain reaction（PCR）or equivalent within the last 72h positive results is available before screening)
4. Hospitalized due to clinical/chest image diagnosis of sever pneumonia. Severe pneumonia defined as dyspnea, hemoglobin oxygen saturation（SpO2）on room air at rest ≤93% or Partial pressure of oxygen（PaO2）/Fraction of inspired oxygen（FiO2）<300 mmHg.

Exclusion Criteria:

1. Subjects who have renal impairment at screening, defined as an estimate glomerular filtration rate (eGFR) <55 ml/min/Body Surface area（BSA）
2. Subjects requiring extracorporeal membrane oxygenation (ECMO) at screening
3. Subjects who are on invasive mechanical ventilator more than 24 hours
4. Female subjects of child-bearing potential (as judged by the Investigator) who do not agree to remain abstinent or use medically acceptable methods of contraception (e.g., implants, injectable, combined oral contraceptives, intra-uterine devices [Intrauterine devices（IUDs）], double-barrier protection) during the study. Male participants who do not agree to use a condom with spermicide during intercourse (if not surgically sterilized) during the study.
5. Subjects who receive anticoagulants overall (except subtherapeutic doses of heparin which is ≤ 6000 International Unit（IU）twice a day Enoxaparin or equivalence) including but not limited to warfarin, rivaroxaban, apixaban, dabigatran acenocoumarol, fencoumarol, or other parenteral anticoagulants at randomization. Antiplatelets drugs are allowed
6. Subjects who have International Normalized ratio or International normalized ratio（INR）>1.3 Upper limit of normal（ULN）.
7. Subjects who have Absolute Neutrophil Count (ANC) <1,000/μL.
8. Subjects who have platelets count <80,000 /μL.
9. Subjects who have activated Partial Thromboplastin Time (aPTT) >1.5 Upper limit of normal（ULN）.
10. Severe anaemia (haemoglobin < 7.0 g/dL).
11. Bleeding in the past 24 hours requiring blood transfusion.
12. Women who are pregnant or lactating at Screening or planning to conceive (self or partner) at any time during the study, including the follow-up period.
13. Subjects who have the following chronic organ dysfunction or immunosuppression:

    1. Heart: New York heart association cardiac function IV.
    2. Lung: severe lung diseases other than COVID-19 lead to home oxygen therapy.
    3. Kidneys: renal impairment requiring chronic dialysis
    4. Liver: liver cirrhosis confirmed by biopsy and clear portal hypertension; the upper digestive tract hemorrhage caused by portal hypertension; or previous liver failure/hepatic encephalopathy/hepatic coma.
    5. Immune function: IV chemotherapy and radiotherapy within 4 weeks before screening or use of immunosuppressive medication within 2 weeks before screening including but not limited to: tacrolimus, cyclosporin, sirolimus, mycophenolate or azathioprine etc., or subjects with leukemia, lymphoma or acquired immunodeficiency syndrome [AIDS].
14. Solid organ or bone marrow transplantation within 4 weeks.
15. The following conditions occurring within 4 weeks prior to screening:

    1. Acute pulmonary embolism
    2. Acute coronary syndrome such as myocardial infarction, unstable angina pectoris etc.
16. Known allergy to the active ingredient of STC3141 or its excipients (i.e., phosphate buffer).
17. The investigator consider participation in the study is not in the best interests of the subjects.
18. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the subject; affect study endpoints or decrease the chance of obtaining satisfactory data required to achieve the objectives of the study.
19. Any other severe or unstable medical condition that, in the opinion of the Investigator or Sponsor, could be expected to progress, recur, or change to such an extent that it could put the subject at special risk, or bias the assessment of the clinical or mental status of the subject to a significant degree.
20. Simultaneous participation in other interventional trials which could interfere with this trial; simultaneous participation in registry and diagnostic trials is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse event（AE）, treatment emergent adverse event（TEAE）, serious adverse event（SAE）, adverse event of special interest（AESI） | up to 30 days

SECONDARY OUTCOMES:
Changes of C-reactive protein（CRP）（mg/dL, or nmol/L, or mg/L） | through study completion, an average of 30 days.
Changes of D-dimer（mg/L, or ng/mL, or μg/mL） | through study completion, an average of 30 days.
Changes of total bleeding time（TBL）（μmol/L） | through study completion, an average of 30 days.
Changes alanine transaminase（ALT）（IU/L, or U/L, or nkat/L） | through study completion, an average of 30 days.
Changes estimated glomerular filtration rate（eGFR）（ml/min） | through study completion, an average of 30 days.
Changes of activated partial thromboplastin time（aPTT）（seconds） | through study completion, an average of 30 days.
Changes of lactate dehydrogenase（LDH）（IU/L, or U/L, or nkat/L） | through study completion, an average of 30 days.
Changes of partial pressure of oxygen（PaO2）/fraction of inspired oxygen（FiO2） ratio | through study completion, an average of 30 days.
Changes of partial pressure of oxygen（PaO2）/fraction of inspired oxygen（FiO2） ratio for subjects who are on invasive or non-invasive ventilator | through study completion, an average of 30 days.
Changes of Sequential Organ Failure Assessment（SOFA）score | through study completion, an average of 30 days.
  Specific score of 0, 1, 2, 3, 4. Higher score indicates worse prognosis.
Time to invasive mechanical ventilation | through study completion, an average of 30 days.
Time to independence from non-invasive mechanical ventilation | through study completion, an average of 30 days.
Time to independence from oxygen therapy | through study completion, an average of 30 days.
Duration of hospitalization | through study completion, an average of 30 days.
All-cause mortality rate | On Day 30.
Subgroup analysis | through study completion, an average of 30 days.

OTHER OUTCOMES:
Changes from baseline in MPO（neutrophil-derived extracellular traps (NETs)）（ng/ml）and citrullinated histone (H3 in plasma)（ng/ml） | up to 7 days
  As an exploratory objective, the change in biomarkers from baseline following STC3141 treatment in subjects with severe COVID-19 pneumonia will be evaluated.
Changes from baseline in interleukin（IL）-1b, interleukin（IL）-2, interleukin（IL）-6, interleukin（IL）-8/CXCL8, interleukin（IL）-10, Interferon（IFN）-γ, tumor necrosis factor（TNF）-α, interleukin（IL）-12/P70（pg/ml） | up to 7 days
  As an exploratory objective, the change in biomarkers from baseline following STC3141 treatment in subjects with severe COVID-19 pneumonia will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: James Pang, PhD, Principal Investigator — Grand Medical Pty Ltd.
Locations (4):
- Belgium (4):
  - Onze-Lieve-Vrouwziekenhuis Aalst, VZW, Aalst
  - Universitair Ziekenhuis Brussel, Brussels
  - Jan Yperman Ziekenhuis vzw, Ieper
  - CHU Liège, Liège

IPD SHARING:
Plan to Share IPD: No